CLINICAL TRIAL: NCT04484805
Title: Continuation of the Development of Moisture Management Liner and Active Cooling System for Improving Residual Limb Skin Care
Brief Title: Socket Cooling Effectiveness Take Home Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Liberating Technologies, Inc. (Industry)
Collaborators: Vivonics, Inc. (Industry)
Responsible Party: Principal Investigator, Todd Farrell, Director of Research, Liberating Technologies, Inc.
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: 120180039; W81XW-17-C-005 (Other: DoD)
Record Dates: First submitted 2020-06-05; First posted 2020-07-24 (Actual); Results first posted 2024-10-22 (Actual); Last update posted 2024-10-22 (Actual); Status verified 2024-10

CONDITIONS: Amputation; Amputation; Traumatic, Leg, Lower; Amputation Stump; Limb; Absence, Congenital, Lower; Prosthesis User; Lower Limb Amputation Below Knee (Injury)
Keywords: cooling; amputee; lower limb absence; prosthesis; prosthetic leg; transtibial; below knee amputation; lower limb difference; lower limb loss; socket; prosthetist; sweat; active; walking; prosthetic liner; prosthetic sock; perspiration; moisture; heat; thermal
MeSH Terms: conditions — Wounds and Injuries; Motor Activity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- ICE Unit (Experimental): The subject wears the experimental socket with an ICE Unit, which includes a TEC and will be actively cooling the leg whenever the device is powered on. An ambient temperature sensor and step counter is attached to the socket. The subject is only informed that each condition is a "different level of cooling" to reduce bias. This condition should last approximately one month.
  Interventions: Device: ICE Condition
- Sham Unit (Sham Comparator): The subject wears the experimental socket with a Sham Unit, which excludes a TEC and will not be actively cooling the leg when the device is powered on. An ambient temperature sensor and step counter is attached to the socket. The subject is only informed that each condition is a "different level of cooling" to reduce bias. This condition should last approximately one month.
  Interventions: Device: Sham Condition

INTERVENTIONS:
Device: ICE Condition — Experimental socket integrated with a heat spreader. An ICE Unit (includes TEC) is attached to the socket.
  Other Names: Cooling Unit; ICE Unit
  Arms: ICE Unit
Device: Sham Condition — Experimental socket integrated with a heat spreader. A Sham Unit (excludes TEC) is attached to the socket.
  Other Names: Sham Unit
  Arms: Sham Unit

SUMMARY:
The comfort and fit of the residual limb within a prosthetic socket are of primary concern for many amputees. The residual limb is typically covered by non-breathable and non- thermally conductive materials that can create a warm and ultimately moist environment.

To address this, Liberating Technologies, Inc. (LTI) and Vivonics, Inc. have developed a thermo-electric cooling (TEC)-based module called the Intrasocket Cooling Element (ICE), that can be embedded into the prosthesis in order to cool the residual limb. A technology that can provide thermal control while retaining adequate suspension, weight and other prosthetic characteristics would benefit many prosthesis wearers.

DETAILED DESCRIPTION:
The comfort and fit of the residual limb within a prosthetic socket are of primary concern for many amputees. The residual limb is typically covered by non-breathable and non- thermally conductive materials that can create a warm and ultimately moist environment. Studies found increases in socket temperature after the prosthesis was donned (0.8 degrees C) and after 30 minutes of walking (2.5 degrees C). Temperatures were found to remain elevated long after activity cessation and even a rest period of double the duration of the preceding activity period is insufficient to return the limb to its initial temperature. A study suggested that a modest temperature increase of only 2 degrees C may be responsible for reports of thermal discomfort by amputees. Therefore, a small amount of activity can cause the socket temperature to elevate and remain at an uncomfortable level for an extended period of time, which can lead to decreased wear times. In summary, an uncomfortable socket/residual limb interface decreases prosthesis use among amputees who want to remain active in their lives.

To address this, Liberating Technologies, Inc. (LTI) and Vivonics, Inc. have developed a thermo-electric cooling (TEC)-based module called the Intrasocket Cooling Element (ICE), that can be embedded into the prosthesis in order to cool the residual limb. A technology that can provide thermal control while retaining adequate suspension, weight and other prosthetic characteristics would benefit many prosthesis wearers.

This study will focus on investigating the efficacy of this novel socket cooling technology.

The rationale for this study is to determine how well the new technology can cool the residual limb not only in a controlled laboratory environment, but also in a home environment where the device would ultimately be utilized.

The primary objective of this study is to measure the effects of cooling the residual limb on quality of life (QoL) and functional outcomes. Cooling the residual limb inside the prosthetic socket would result in less sweating and greater comfort while wearing the prosthesis, and ultimately greater function and better quality of life as measured by standard functional and QoL outcome measures.

A two group, prospective, double-blinded, block randomized, crossover study design will be implemented. Research participants will be consented and have baseline activity and socket temperature data collected from their usual prosthesis during normal use (4 weeks). The ICE system will be integrated into a custom, experimental socket for each subject. Two versions of the cooling module will be created: (1) a fully-functional, active ICE cooling module (the so called "ON", or experimental, condition), and (2) a placebo ICE module with the TEC unit replaced with an insulating material layer between the fan and the heat spreader such that even when the system is turned on, minimal heat transfer occurs (the control, or "OFF" condition). An ICE module with a heat spreader will be embedded into the socket and the fan will continue to run whether or not active cooling is engaged for both test conditions; however, no heat will be able to be transferred through the insulating layer in the OFF condition. The TEC inside the ICE unit will not be visible once assembled and the modules will be assembled independently; therefore, both the subject and the tester will be blinded to the condition being tested for both the in-lab and at-home testing. A serial number will be used to identify the assembled units and the master key stored separately.

The participants will be divided into two groups and the order of the experimental conditions will be randomized. Each condition will be tested for 4 weeks. In-lab testing and functional measures will be assessed between testing periods as additional assessments of efficacy of the device. Testing will consist of 4 test site visits, as well as 1-2 visits to create and align the experimental socket. The entire study will continue for 3 months.

Lower limb prosthesis users will be recruited for the study and consented with an approved protocol. Research participants will represent a convenience sample and will reflect the local population of both above-knee (AK) and below-knee (BK) amputees of various K-levels using a variety of suspension types who could benefit from temperature control within the socket.

A maximum of 20 subjects will be recruited for this study. This is increased from the target 16 subjects to account for any drop-outs, etc.

ELIGIBILITY:
Inclusion Criteria:

* Must have a lower limb absence
* Willing and able to complete outlined tasks
* Must complete and pass our Semmes-Weinstein monofilament test
* Must understand English in order to be properly consented and provide feedback to the study personnel

Exclusion Criteria:

* The risks to pregnant women and fetuses are unknown and therefore pregnant women should not participate in the study
* No symptoms consistent with peripheral neuropathy or other sensory diagnosis that could prevent them from feeling the temperature of their limb

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2020-11-03 (Actual); Study Completion 2020-11-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Liberating Technologies, Inc., Holliston, Massachusetts
  - Minneapolis VA, Minneapolis, Minnesota

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- ICE Unit First, Then Sham Unit: The subject wears the experimental socket with an ICE Unit, which includes a TEC and will be actively cooling the leg whenever the device is powered on. An ambient temperature sensor and step counter is attached to the socket. The subject is only informed that each condition is a "different level of cooling" to reduce bias. This condition should last approximately one month.
  The subject is then swapped to the Sham condition, which is the same setup as above except it excludes a TEC and will not be actively cooling the leg when the device is powered on. They will be in this condition for approximately one month.
  ICE Condition: Experimental socket integrated with a heat spreader. An ICE Unit (includes TEC) is attached to the socket.
  Sham Condition: Experimental socket integrated with a heat spreader. A Sham Unit (excludes TEC) is attached to the socket.
- Sham Unit First, Then ICE Unit: The subject wears the experimental socket with a Sham Unit, which excludes a TEC and will not be actively cooling the leg when the device is powered on. An ambient temperature sensor and step counter is attached to the socket. The subject is only informed that each condition is a "different level of cooling" to reduce bias. This condition should last approximately one month.
  The subject is then swapped to the ICE condition, which is the same setup as above except it includes a TEC and will be actively cooling the leg when the device is powered on. They will be in this condition for approximately one month.
  ICE Condition: Experimental socket integrated with a heat spreader. An ICE Unit (includes TEC) is attached to the socket.
  Sham Condition: Experimental socket integrated with a heat spreader. A Sham Unit (excludes TEC) is attached to the socket.
Period: Overall Study
Arm/Group | ICE Unit First, Then Sham Unit | Sham Unit First, Then ICE Unit
Started | 6 | 6
Completed | 4 | 6
Not Completed | 2 | 0
Not completed — LTI_H01 piloted the device and was too familiar with the study design to be unblinded/analyzed | 1 | 0
Not completed — LTI_H02 had socket fit issues causing discomfort which caused us to withdraw them from the study. | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- ICE Unit, Then Sham Unit: The subject wears the experimental socket with an ICE Unit, which includes a TEC and will be actively cooling the leg whenever the device is powered on. An ambient temperature sensor and step counter is attached to the socket. The subject is only informed that each condition is a "different level of cooling" to reduce bias. This condition should last approximately one month.
  The subject is then swapped to the Sham condition, which is the same setup as above except it excludes a TEC and will not be actively cooling the leg when the device is powered on. They will be in this condition for approximately one month.
  ICE Condition: Experimental socket integrated with a heat spreader. An ICE Unit (includes TEC) is attached to the socket.
  Sham Condition: Experimental socket integrated with a heat spreader. A Sham Unit (excludes TEC) is attached to the socket.
- Sham Unit, Then ICE Unit: The subject wears the experimental socket with a Sham Unit, which excludes a TEC and will not be actively cooling the leg when the device is powered on. An ambient temperature sensor and step counter is attached to the socket. The subject is only informed that each condition is a "different level of cooling" to reduce bias. This condition should last approximately one month.
  The subject is then swapped to the ICE condition, which is the same setup as above except it includes a TEC and will be actively cooling the leg when the device is powered on. They will be in this condition for approximately one month.
  ICE Condition: Experimental socket integrated with a heat spreader. An ICE Unit (includes TEC) is attached to the socket.
  Sham Condition: Experimental socket integrated with a heat spreader. A Sham Unit (excludes TEC) is attached to the socket.
- Total: Total of all reporting groups
Arm/Group | ICE Unit, Then Sham Unit | Sham Unit, Then ICE Unit | Total
Number analyzed (Participants) | 6 | 6 | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 5 | 9
  >=65 years | 2 | 1 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 5 | 6 | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 6 | 6 | 12
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 6 | 6 | 12

OUTCOME MEASURES:

1. Primary Outcome: Residual Limb Temperature
Description: This will be tested only during in-lab visits. An intervention of the experimental socket with the ICE cooling unit should yield at least a 2 degree Celsius decrease in temperature compared with no intervention. This will be tested in-lab with 6 thermocouples taped to the residual limb while the subject is sitting and walking on a treadmill.
  The reported result is the temperature difference of the residual limb from the baseline temperature (before activity) to the end of the sitting period (after activity). The ICE or Sham unit is turned on 5 minutes before the 15 minute walking period. After the 15 minute walking period, the participant sits with the unit ON for 45 minutes. The baseline temperature reading is taken directly before the unit is turned on, and the end temperature reading is taken after the 45 minutes of sitting.
Time Frame: 4 hours
Measure: Mean (Standard Deviation); unit: Avg Temp Diff from Baseline (Degrees C)
Arm/Group | ICE Unit | Sham Unit
Number analyzed (Participants) | 12 | 12
Avg Temp Diff from Baseline (Degrees C) | -2.3 (0.9) | 1.9 (2.0)

ADVERSE EVENTS:
Time Frame: Adverse events were monitored/collected during the experimental conditions. With each condition lasting about 1 month, each participant was monitored for adverse events for about 2 months. Adverse events were monitored/assessed at least every 2 weeks by phone call, with study staff checking in more frequently if participants reached out with questions. Participants were told to reach out to study staff immediately if adverse events did occur.
Arm/Group | ICE Unit | Sham Unit
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 0/12 | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2019-07-12): https://cdn.clinicaltrials.gov/large-docs/05/NCT04484805/Prot_001.pdf